CLINICAL TRIAL: NCT06988410
Title: Unstable Income, Rising Stress? The Effect of Income Instability on Psychological and Physiological Health
Brief Title: Income Volatility and Mental Health, Full Experiment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OSP169128; R01AG076655 (NIH)
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Depression; Anxiety; Blood Pressure
Keywords: income instability; uncertainty
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): The Control arm will not be hired by the cash-for-work program but will be surveyed.
- Stable Income Arm (Experimental): The Stable Income arm will work the same amount and earn the same amount every period.
  Interventions: Behavioral: Work opportunities
- Predictable Instability Arm (Experimental): The hours and earnings of the Predictable Instability arm will vary over time. In three periods, the participant will work longer hours and will earn more. In the remaining three periods, she will work fewer hours and will earn less. However, on average, the work offered will be the same as in the stable arm. Crucially, she will be able to predict all swings in her study earnings in the future-i.e., she will know her hours and earnings in each future period.
  Interventions: Behavioral: Work opportunities
- Unpredictable Instability Arm (Experimental): The hours and earnings of the Unpredictable Instability arm will vary unpredictably over time. In any given period, there will be a 50% chance that she works longer hours and earns more and a 50% chance that she works fewer hours and earns less. The expected average earnings remain the same as the stable arm and the predictable arm, though specific individuals may earn more or less.
  Interventions: Behavioral: Work opportunities

INTERVENTIONS:
Behavioral: Work opportunities — Individuals in the treated arms of the study will be offered work opportunities (sewing bags) to earn cash. The timing of these opportunities and knowledge of the amount and timing varies by experimental arm.
  Arms: Predictable Instability Arm; Stable Income Arm; Unpredictable Instability Arm

SUMMARY:
Income instability is a defining aspect of the lives of the poor, who also disproportionately suffer from poor mental and physical health. This research is the first to assess the causal effects of predictable and unpredictable income instability on the psychological and physical health of the poor. It will advance the scientific knowledge on the effects of economic instability as well as understanding of health gaps across populations.

DETAILED DESCRIPTION:
The poor suffer disproportionally from poor mental and physical health. Many causes for these differences have been considered, including low income. But, poor families' incomes are not only low, but also often unstable and unpredictable. This instability creates uncertainty about whether individuals will be able to safeguard their future well-being. According to the allostatic load framework, prolonged activation of physiological stress responses will cause "wear and tear" on the body, heightening risks of cardiovascular disease and of age-related metabolic diseases, promoting cognitive decline and dementia, and accelerating cellular aging.

This research will study the causal effects of income instability on the psychological and physical health of the poor. The study's specific aims are to: 1) Identify the causal effect of income instability on psychological health (e.g. depression, anxiety), and physical health (e.g. blood pressure), 2) Decompose the effects identified in aim 1 into the effects of predictable and unpredictable instability and compare to the impact of increasing the average level of income, and 3) Investigate the channels through which effects on health occur, including both economic and behavioral channels and estimate the impact of key moderating factors (e.g. age, baseline mental health).

The trial will be conducted in northern Ghana. It will manipulate income instability by varying the number of work hours (and hence earnings) of participants in a cash-for-work program. Participants in the first treatment arm will have a fixed work schedule, with the same hours and earning each period. The hours and earnings of a second treatment arm will vary over time, but the fluctuations will be known in advance. Finally, the number of work hours and earnings of a third treatment arm will fluctuate unpredictably. Each of these arms will be compared to a control group that is surveyed, but not offered additional work. Importantly, the study will vary income instability while holding the average level of income constant in order to disentangle the impact of instability from the level-effect.

The study will create 1,867 new jobs that would not otherwise be available during the lean season when jobs are scarce. The intervention has been designed so that the job opportunity cannot make the participants worse off than they would otherwise have been in the absence of research.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18 - 60
* Female
* Lives in a household with 5 or fewer adults

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2267 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-10-12 (Estimated)

PRIMARY OUTCOMES:
Depression | The measurement will be taken at endline (after 6 2-week periods of intervention). Respondents will be asked to evaluate each item over the last 10 days.
  Patient Health Questionnaire (PHQ)-8, each item is scored 0-3. Multiplying the range per item (0-3) by the number of items (8) gives the total corresponding range of the scale: 0 to 24. Higher scores indicate worse mental health.
Anxiety | The measurement will be taken at endline (after 6 2-week periods of intervention). Respondents will be asked to evaluate each item over the last 10 days.
  Generalized Anxiety Disorder (GAD)-7 scale, each item is scored 0-3. Multiplying the range per item (0-3) by the number of items (7) gives the total corresponding range of the scale: 0 to 21. Higher scores indicate worse mental health.
Dietary Diversity | The measurement will be taken at endline (after 6 2-week periods of intervention). Respondents will be asked to evaluate each item over the last ten days.
  The Household Dietary Diversity Score is used to measure households' food access on the number of food groups they had consumed (out of 11). The measure sums the number of categories with any positive consumption by the household resulting in a total score between 0 and 11. Households that consume a greater number of food groups are considered to have greater dietary diversity (i.e. more is better).
Blood Pressure | The measurement will be taken at endline (after 6 2-week periods of intervention).
  Blood Pressure Measurement, recorded in millimeters of mercury (mmHg) with two components: systolic and diastolic. Higher values indicate increased cardiovascular risk

CONTACTS AND LOCATIONS:
Locations (1):
- Innovations for Poverty Action, Tamale, Ghana

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD collected throughout the study
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Within 1 year after publication with no end date
Access Criteria: No criteria, any individual who would like to download it from the PI's website or a public repository.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT06988410/ICF_000.pdf